CLINICAL TRIAL: NCT06662604
Title: Evaluation of Bone Marrow Stem Cells Concentrate with Platelet Rich Fibrin and Bone Graft in Bone Regeneration of Maxillary Cystic Defects Versus Platelet Rich Fibrin with Bone Graft (a Randomized Controlled Trial)
Brief Title: Using of Bone Marrow Stem Cell Concentrate with Platelet Rich Fibrin and Bone Graft in Bone Reconstruction of Upper Jaw Bony Cystic Defects, Comparing with Platelet Rich Fibrin with Bone Graft
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Motea Abdulsalam Sanad, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMFS 3-3-18
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Maxillary Cyst
Keywords: maxillary cyst; bone marrow stem cells; platelet rich fibrin PRF; bone graft; bone reconstruction; jaw cyst
MeSH Terms: conditions — Jaw Cysts | interventions — Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Stem cells ,PRF group) intervention group (Experimental)
  Interventions: Biological: Bone marrow stem cells concentrate , platelet rich fibrin , bone graft
- Group B (PRF group) (Active Comparator)
  Interventions: Biological: platelet rich fibrin and bone graft

INTERVENTIONS:
Biological: Bone marrow stem cells concentrate , platelet rich fibrin , bone graft — All participants will be treated with Bone marrow stem cells concentrate , platelet rich fibrin , bone graft.
  Arms: Group A (Stem cells ,PRF group) intervention group
Biological: platelet rich fibrin and bone graft — All participants will treated with platelet rich fibrin PRF , bone graft.
  Arms: Group B (PRF group)

SUMMARY:
Will the use of bone marrow stem cells with platelet rich fibrin enhance and accelerate the bone regeneration in the upper jaw cystic defects ?

DETAILED DESCRIPTION:
Reconstruction of critical size bone defect in maxillofacial surgery is a great challenge, current practice of bone reconstruction still having problems like delay in bone regeneration (up to 12 months) and bone graft failure and low availability of autogenous bone graft.

last decade stem cells therapy gained great interest, in many studies Bone marrow stem cells showed promising result in bone regeneration enhancing .

Platelet Rich Fibrin PRF also capability of enhancing bone and tissue regeneration by releasing of certain protein molecules call growth factors that initiate sequential biological events resulting in stem cells migration into the site of bone defect and differentiation to bone formation cells (osteoblast cells ).

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-50 years
* Patients with a critical size maxillary cyst. (>3 cm)
* Patients that free of any significant medical conditions that could affect healing or outcomes.

Exclusion Criteria:

* Patients with large jaw cyst that endanger vital structures
* Patients with significant medical condition
* age under 18 years

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-10-26 (Estimated); Primary Completion 2025-09-17 (Estimated); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
cyst volume | preoperative and 3, 6 months postoperative.
  volumetric analysis of cystic defect 3, 6 months after treatment .

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu M, Liu Y, Luo F. The role and mechanism of platelet-rich fibrin in alveolar bone regeneration. Biomed Pharmacother. 2023 Dec;168:115795. doi: 10.1016/j.biopha.2023.115795. Epub 2023 Nov 2. PMID 37918253
- [Background] Matsumura-Matsuo M, To M, Okudera T, Matsuo M. Regeneration processes of alveolar bone and microvascular changes after the application of platelet-rich fibrin. J Oral Biosci. 2023 Sep;65(3):218-225. doi: 10.1016/j.job.2023.05.004. Epub 2023 Jun 3. PMID 37277026
- [Background] Fitzsimmons REB, Mazurek MS, Soos A, Simmons CA. Mesenchymal Stromal/Stem Cells in Regenerative Medicine and Tissue Engineering. Stem Cells Int. 2018 Aug 19;2018:8031718. doi: 10.1155/2018/8031718. eCollection 2018. PMID 30210552
- [Background] Manfrini M, Di Bona C, Canella A, Lucarelli E, Pellati A, D'Agostino A, Barbanti-Brodano G, Tognon M. Mesenchymal stem cells from patients to assay bone graft substitutes. J Cell Physiol. 2013 Jun;228(6):1229-37. doi: 10.1002/jcp.24276. PMID 23129455
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31799249/